CLINICAL TRIAL: NCT01836393
Title: Efficacy Study on Symptomatic Control of Patient With Knee Osteoarthritis Between 14% of Plai (Plaivana®) to Placebo Gels
Acronym: OA knee Plai
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: and Bangkok drugs Co. (Unknown)
Responsible Party: Principal Investigator, Weerachai Kosuwon, Department of Orthopedics, Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KKU Ortho Plai
Record Dates: First submitted 2013-04-09; First posted 2013-04-19 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Knee Osteoarthritis
Keywords: Plai; Efficacy; OA knee; The efficacy study of Plai cream for OA knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- placebo and plai (Experimental): The essential plai cream has anti-inflammatory and antimicrobial effects (Wasuwat1989, Giwanon 2000, Pithayanukul 2007, and Tripathi 2008). Active chemicals of plai cream are composed of sabinene, alpha and gamma tepinenes, terpinen 4-ol and (E)-1-(3,4-dimethoxyphenyl butadiene (DMPBD). The DMPBD has a property of anti-inflammatory activity(Ozaki 1991, Jeenapongsa 2003). Plavina® 40 mg in 100 gm (contains DMPBD of …%). This product was supplied in lacquered aluminum collapsible tube containing 100 gram cream packing.
  Interventions: Drug: Plavina cream

INTERVENTIONS:
Drug: Plavina cream — The essential plai cream has anti-inflammatory and antimicrobial effects (Wasuwat1989, Giwanon 2000, Pithayanukul 2007, and Tripathi 2008). Active chemicals of plai cream are composed of sabinene, alpha and gamma tepinenes, terpinen 4-ol and (E)-1-(3,4-dimethoxyphenyl butadiene (DMPBD). The DMPBD has a property of anti-inflammatory activity(Ozaki 1991, Jeenapongsa 2003). Plavina® 40 mg in 100 gm (contains DMPBD of …%). This product was supplied in lacquered aluminum collapsible tube containing 100 gram cream packing.

SUMMARY:
To determine whether plai cream is effective in treating mild to moderate degrees of osteoarthritis of the knee in the elderly patient compared with placebo cream.

DETAILED DESCRIPTION:
Osteoarthritis is the most common of the arthritides, affecting at least 20 million Americans, a number that is expected to double over the next two decades. currently available medical therapies primarily address the treatment of joint pain in patients with osteoarthritis.Analgesics as well as traditional and cyclooxygenase-2-selective nonsteriodal anti-inflammatory drugs (NSAIDs) have suboptimal effectiveness,and there is some question about their safety, especially in the light of recent reports of increased cardiovascular risk.

Plai (Zingiber cassumunar Roxb.) belongs to family of Ginger. Plai essential cream also has an activity on scavenging H2O2 generated by ultrasound exposure. The dilutions of 1:2,000 and 1:1,000 (v:v) of plai cream presented H2O2 scavenging activity by reducing emissions of DCFH-fluorescence within U937 cells, compared with the cell control. Plai essential cream inhibited nitric oxide (NO) production in the macrophage cell line (J774), compared with untreated cells. However, high concentrations of plai cream (1:1 and 1:10), were toxic to U937 and J744 cell lines. Moreover, plai cream at dilutions of 1:1,000 and 1:2,000, significantly inhibited COX II activity in treated cells compared to the untreated cells. Three major compounds of plai essential cream were sabinene, terpinen-4-ol and (E)-1-(3,4-dimethyoxyphenyl) butadiene respectively.There have been many studies on the efficacy of Plai as an analgesic and anti-inflammatory when applied directly to the affected area. The majority of these studies have been carried out in Thailand as this is where the plant originates from and it is used extensively in Thai massage and herbal medicine. The anti-inflammatory activity of a compound found in Plai extracts was assessed and compared with aspirin, and two other lesser known anti-inflammatory drugs. The results obtained showed that the anti-inflammatory effect of the compound (compound D) mainly occurred in the acute phase of inflammation.Moreover, the anti-inflammatory affect of plai oil was twice as potent as Diclofenac. The Plai cream was shown to reduce swelling and pain significantly in athletic ankle sprain in the first 2-3 days of the treatment.

These findings suggest that topical plai cream is a safe and potentially useful drug for the treatment of painful OA of the joints, however, there has been no efficacious study on the plai cream namely Plaivana® for relieving symptoms in patient with OA knee joint before, therefore, this study is proposed.

Subject selection and withdrawal criteria Number of subjects A sufficient number of subjects with OA of the knee will be screened in order to randomize at least 100 subjects (100 pairs) The study should provide 92 subjects (92 pairs) evaluable subjects, assuming that 10% of subjects will withdraw before having one the last assessment in the primary outcome variable.

Objectives Primary To evaluate the pain control using VAS of Plai cream 14 gm/100 (Plaivana®) compared with placebo cream in patient with OA knee.

Secondary

* To evaluate the WOMAC score of patients in the Plaivana® compared with the placebo groups.
* To compare the amount of acetaminophen tablet taking in both groups.
* To compare the side effect of Plaivana® with the placebo. Investigational plane Study Design This will be the phase III randomized, double-blind, placebo-controlled cross-over trial of 12 weeks duration. This study is designed to evaluate the efficacy of Plaivana® to placebo, in adults with OA of the knee. Randomization will be stratified by Kellgren-Lawrence (KL) grading (grade 2 and 3) using X-ray standing MTP technique. A total of 100 subjects (100 pairs of subjects) are planned for enrollment in this study. This study will be conducted over approximately 12 weeks.

Patients and Methods Patients and study design This was the phase III randomized, double-blind, placebo-controlled cross-over trial of 12 weeks duration designed to evaluate the efficacy of Plaivana® to placebo, in adult with OA of the knee. A total of 100 subjects (100 pairs of subjects) are planned for enrollment in this study. This was an 8 weeks period of study treatment-control periods (4 weeks for treatment, two weeks for wash-out and 4 weeks for placebo periods). The study was conducted in accordance with the Declaration of Helsinki, was approved by Khon Kaen University Ethics Committee for Human Research and informed consent was obtained from all patients.

Study medication The essential plai cream has anti-inflammatory and antimicrobial effects (Wasuwat1989, Giwanon 2000, Pithayanukul 2007, and Tripathi 2008). Active chemicals of plai cream are composed of sabinene, alpha and gamma tepinenes, terpinen 4-ol and (E)-1-(3,4-dimethoxyphenyl butadiene (DMPBD). The DMPBD has a property of anti-inflammatory activity(Ozaki 1991, Jeenapongsa 2003). Plavina® 40 mg in 100 gm (contains DMPBD of …%). This product was supplied in lacquered aluminum collapsible tube containing 100 gram cream packing.

Treatment Assignment and dosing Subjects will be assigned to study treatment in accordance with the randomization schedule. Randomization will be stratified by KL grade (grade 2 or 3). At the Baseline/Randomization Visit, each subject will be randomly assigned to either Plaivana® or placebo creams. Plaivana® or placebo creams were applied three times around the index knee. The 2 inches in length of cream was topically applied to the skin around the index knee joint, then rubbing the cream until it dry. After applying the cream, patients should wash their hands and do not touch their eyes.

Blinding This is a double-blind study. All study drugs will be blinded to the investigators and subjects. The study and placebo creams were prepared in the same lacquered aluminum collapsible tube containing 100 gram cream packing.

Product Accountability In accordance with the standard requirements, the investigator must document the amount of investigational cream product dispensed and /or administered to study returned to the investigator. Product accountability records must be maintained throughout the course of the study.

Treatment Compliance A drug-dispensing log will be maintained by the investigator. Subjects will be instructed at the baseline visit to record the dates on which they applied the cream from each lacquered aluminum collapsible tube and to bring the tube with them on study visit days. Subject compliance will be assessed based on the weight of returning tube, which will be collected and recorded in the Data Record Form. Subject will be asked to complete a diary card to capture daily applying doses of the cream.

Concomitant Medications and Non-drug therapies Subject was asked to complete a diary card to capture daily applying doses of the cream. Subject was asked to complete a diary to capture takes and changes in concomitant therapy during the study, including pain medication or nutritional supplements for OA related pain. Subjects were permitted to take acetaminophen (500 mg) three times or two tablets for pain every 4-6 hours. Other topical analgesics, NSAID and COX-2 inhibitors are prohibiting. All concomitant medications or nutritional supplement taken during the study were also recorded.

During wash-out period Subjects were permitted to take only acetaminophen for OA pain for 7 days. Subjects maintained written diaries to record dosing of medications and nutritional supplements for OA-associated pain.

STUDY ASSESSMENT AND PROCEDURES Subjects will be expected to attend the clinic a minimum of 6 times over period of approximately 12 weeks. The study consists of 7 phases: screen, treatment, follow-up, washout, screening, treatment, and follow-up.

The study investigation will discuss with each subject in detail of the study objectives, its requirement and its restrictions.

The screening 1st visit will include a formal review of the complete medical history, all concurrent medications, concomitant diseases, medication taken within the last month and all medications of interested in the exclusion criteria, and other eligibility requirement for the study including contraindication for plai cream.

Eligible subject will further be determined by exclusion criteria such as severe pain defined as above 80 mm on the 100 mm VAS scale for pain, as identified by subject response to WOMAC pain subscale.

If OA present in both knees the investigator will identify which knee will be X-ray for the study entry, with preference for the knee with more severe pain (<80 mm on WOMAC pain sub scale) A radiograph of the index knee will be obtained using the MTP technique to evaluate JSW and KL grade. The minimum JSW must be at least 1.5 mm in the medial compartment and at least 2.5 mm in the corresponding lateral compartment with KL grade of 2 or 3.

At the screening 1st visit, subject should be instructed to withhold OA medication for pain for 7 days for all NSAIDs or 24 hours for acetaminophen immediately prior to the baseline visit.

At the 2nd visit subject will be randomized following stratification by KL grade. This visit, the following procedures will be completed:

* VAS
* WOMAC Subject will be received their first study or placebo cream, acetaminophen 500 mg for 40 tablets and daily record their symptoms.

Efficacy Assessments Primary endpoint VAS: The primary endpoint is the change from baseline in VAS. This endpoint will be measured at visit 2-13 (week 1-12) Secondary endpoint WOMAC Score The WOMAC score is a tri-dimensional, disease-specific, self-administered health status measure, probing clinically important, subject-relevant symptoms in the area of pain. The subject will answer WOMAC question on pain subscale, using the Linkert scale 0-100 at screening 1st visit to determine eligibility for inclusion in the study. The subject will complete the entire WOMAC questionnaire during visit 2-13 (week 1-12) Safety Assessments Adverse events The investigator will be responsible for detecting, documenting and reporting events that meet the definition of adverse events. Definition of an adverse event is any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding, for example; skin rash, swelling), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered as an adverse event.Any adverse event should be documented on the patient chart and reported on the Adverse Event Form.

Dropouts Reason for dropout The patients may drop-out of the study if they decide to do so, at any time and irrespective of the reason, or this may be the investigator decision. All dropouts must be documented and the investigator must give the reason.

Data Analysis and statistical considerations Sample size determination The primary endpoint was the change from baseline in visual analog scale (VAS).The secondary endpoint was the Western Ontario McMaster score (WOMAC). These endpoints were measured every week for 9 weeks (4 weeks for each treatment periods and one week for washout period). This study is determined to demonstrate that Plaivana® is able to reduce the pain (VAS), functional score and stiffness score when compared to placebo cream. It is expected that Plaivana® will reduce the VAS by 1.23 (which considers Minimal Clinical Improvement Important, MCII) and SD was 4.39. The significant level is 95% or alpha at 5% of two-sided test and power for detecting different is 80% or beta at 20%. Therefore, the sample size of 103 pairs of patient is needed. Adding 5% dropout rate, we would need approximately 108 pairs of patient (108 patients) to be randomized to each treatment group in the study.

N pairs = ½(1+1/λ)[(Z1-α/2+Z1-β)2/D2pair +( Z2 1-α/2)/2] Λ= number of controls:case = 1 D= Effect size =VAS difference/SDof VAS The VAS difference which minimal clinical improvement important was 1.23 and SDof VAS = 4.39, therefore the sample size was 103 pairs Hypothesis testing The null hypothesis to be tested is that the VAS in Plaivana® group is not different from the placebo group.

Analysis population The primary analysis will be based on patients on intent-to-treat (ITT) population, which will include all patients with baseline results of VAS, WOMAC score.

Statistic methods The mean different of VAS in Plaivana® and placebo be analyzed by Z test, 95% CI of the mean different of VAS. The confident interval of the mean of VAS in each treatment group will be calculated. Other baseline factors such as WOMAC, Stiffness score and acetaminophen used will be analyses by ANOVA, student T test and Mc Nemar 's Chi-square. All statistical analyses were performed by using STATA Statistical Software: Release 10th. (StataCorp. 2007. Stata Statistical Software: Release 10th. College Station, TX: SataCorp.) Data Management The data collection will be done by research assistance using the DATA RECORD FORM SHEATH. Clinical data management will perform in according with the Good Clinical Practice Guidelines.

Ethics The trial will be considered in accordance with: The Declaration of Helsinki adopted by the World Medical Assembly in June 1964, amended at Tokyo in October 1975, at Venice in October 1983 at Hong Kong in September 1989 and at Somerset West in October 1996.

Before a subject included in the trial, the aims and methods of the trial are explained to the subject. The subject givens his/her consent in writing on an information and informed consent form. The investigator will submit the documents required by the regulations according to the Ethics Committee of Khon Kaen University and will obtain their opinion in writing. Subjects cannot be included until the approval of the Ethics Committee has been received.

Quality control-Quality assurance The investigator in charge of the study ensures the efficient organization and good quality of the study, notably he is responsible for protocol compliance, data collection and Good Clinical Practice in general. Data collection will be monitored throughout the study by the monitors after quality control by the investigator.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study met all of the following criteria:

1. Subjects who are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Ambulatory nom pregnant females and males 40-<80 years of age.
3. Subjects who withdraw pain medication or nutritional supplements for symptom relief for knee OA for a total of at least 15 days before screening.
4. Pain at or below 80 mm on a 100 mm VAS in the index knee.
5. A documented diagnosis of OA of the knee, or meeting American College of Rheumatology (ACR) clinical criteria for classification of idiopathic (primary) OA for at least 6 months prior to screening. If OA is presented in both knees the investigator will identify which knee will be X-rayed for study entry, with preference for the knee with more severe pain (<80mm VAS).
6. Has documented radiographic evidence of OA of the knee from the screening Visit radiograph of grade 2 or 3 according to Kellgren and Lawrence Radiographic Grading (11)
7. Subjects with baseline minimum joint space width in the medial and lateral compartments of the index knee of > 1.5 mm and > 2.5 mm at Baseline respectively, measured from radiographs using the MTP view.

Exclusion Criteria

Subjects with any of the following criteria must not be enrolled in the study:

1. Subjects with history of hypersensitivity to Plai.
2. Subjects with skin lesion at the index knee.
3. A history of lower extremity surgery within 6 months prior to screening.
4. Significant prior injury to the index knee within 12 months prior to screening
5. Disease of the spine or other lower extremity joints of sufficient degree to affect the index knee.
6. Treatment with other drugs potentially affecting bone or cartilage metabolism as described below:

   * chronic systematic corticosteroids
   * hyaluronan injection into the index knee with in the previous 6 months.
   * Diacerin or Glucosamine treatment within the last 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
This endpoint will be VAS, measured at visit 2-13 (week 1-12) Primary endpoint VAS: The primary endpoint is the change from baseline in VAS. This endpoint will be measured at visit 2-13 (week 1-12) VAS | 3 months
  VAS 0-100 mm. using questionnaire

SECONDARY OUTCOMES:
WOMAC and | 3 months
  The WOMAC score is a tri-dimensional, disease-specific, self-administered health status measure, probing clinically important, subject-relevant symptoms in the area of pain. The subject will answer WOMAC question on pain subscale, using the Linkert scale 0-100 at screening 1st visit to determine eligibility for inclusion in the study. The subject will complete the entire WOMAC questionnaire during visit 2-13 (week 1-12)

CONTACTS AND LOCATIONS:
Overall Officials: Weerachai Kosuwon, Doctor, Principal Investigator — Department of Orthopedics, Faculty of Medicine, Khon Kaen University, Thailand
Locations (2):
- Thailand (2):
  - Department of Orthopedics, Faculty of Medicine, Khon Kaen University, Thailand, Khon Kaen, Changwat Khon Kaen
  - Faculty of Medicine KhonKaen University, Khonkaen, KhonKaen

REFERENCES:
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Murray CJ, Lopez AD. Mortality by cause for eight regions of the world: Global Burden of Disease Study. Lancet. 1997 May 3;349(9061):1269-76. doi: 10.1016/S0140-6736(96)07493-4. PMID 9142060
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] Ozaki Y, Kawahara N, Harada M. Anti-inflammatory effect of Zingiber cassumunar Roxb. and its active principles. Chem Pharm Bull (Tokyo). 1991 Sep;39(9):2353-6. doi: 10.1248/cpb.39.2353. PMID 1804548
- [Background] Nakatani N. Phenolic antioxidants from herbs and spices. Biofactors. 2000;13(1-4):141-6. doi: 10.1002/biof.5520130123. PMID 11237173
- [Background] Guccione AA, Felson DT, Anderson JJ, Anthony JM, Zhang Y, Wilson PW, Kelly-Hayes M, Wolf PA, Kreger BE, Kannel WB. The effects of specific medical conditions on the functional limitations of elders in the Framingham Study. Am J Public Health. 1994 Mar;84(3):351-8. doi: 10.2105/ajph.84.3.351. PMID 8129049